CLINICAL TRIAL: NCT05725746
Title: Enhancing Cardiovascular Health Equity in Mothers and Children Through Home Visiting
Brief Title: Feasibility of Remote Data Collection With a Point of Care Device to Measure HbA1c
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 202212059
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Pregnant; Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Point of care device to measure HbA1c — After consent the participant will meet with the research team virtually to obtain HbA1c. The HbA1c self check equipment will be sent to the participant. During the video call the research team will talk the participant through obtaining their HbA1c with the point of care device.
  Other Names: A1C Now self check

SUMMARY:
Conduct a pilot study to test feasibility of doing remote data collection with a point of care device that measures HbA1c.

DETAILED DESCRIPTION:
The foundation for cardiovascular health (CVH) is laid in early life by intergenerational interactions, passed from parent to child, that have long-lasting biological and behavioral consequences. Lifestyle interventions can promote CVH among mothers and their children over time. Academic partnerships with home visiting organizations that reach families experiencing health disparities advance intergenerational CVH equity. For this pilot study we are testing the feasibility of doing remote data collection with a point of care device that measures HbA1c to use in the main study.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Screened or participating in NCT04253977
* Able to give informed consent for participation

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For the participants only women will be included: Including only female participants is scientifically justified, as the main study focus is addressing cardiovascular health of prenatal and postpartum women.
Study Population: Pregnant or postpartum women who are currently or have recently participated in the Parents as Teachers home visiting program.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Haire-Joshu, PhD, Principal Investigator — Washington University School of Medicine; Victor G Davila-Roman, MD,FACC,FASE, Principal Investigator — Washington University School of Medicine; Rachel G Tabak, PhD, RD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Only data with identifiers removed will be shared publicly. Any identified data to be shared will only be done so in coordination with the Human Research Protection Office at Washington University in St. Louis and the Institutional Review Board (IRB) at the requesting investigator's institution.
  Datasets with identifiers will only be accessible to study team members with appropriate Human Subjects training.

RESULTS

PARTICIPANT FLOW:
Groups:
- Point of Care Device: Test the feasibility of doing remote data collection with a point of care device that measures HbA1c.
Period: Overall Study
Arm/Group | Point of Care Device
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Point of Care Device
Number analyzed (Participants) | 18
Age, Continuous [Mean (Full Range); unit: Years] | 30 [19 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Feasibility to Obtain HbA1c Through Remote Data Collection
Description: Feasibility will be measured by how many participants are able to obtain HbA1c measure through remote data collection and participant's satisfaction with this means of data collection.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Point of Care Device
Number analyzed (Participants) | 18
Participants
  Able to use point of care device | 17
  Agreed or strongly agreed instructions were helpful | 16

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the data collection visit, about 20 minutes.
Groups:
- Point of Care Device: Participants were asked to test the feasibility and rate the acceptability of using the point of care device.
Arm/Group | Point of Care Device
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/46/NCT05725746/Prot_ICF_000.pdf